CLINICAL TRIAL: NCT02105311
Title: A Prospective, Randomized Study Comparing the Effects of Selective Laser Trabeculoplasty and Travoprost on the Circadian Intraocular Pressure Variation
Brief Title: Effect of Selective Laser Trabeculoplasty Versus Travoprost on Circardian Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Weerawat Kiddee, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC57-020-02-1
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Intraocular Pressure
Keywords: Intraocular pressure; Selective laser trabeculoplasty; Travoprost; Ocular surface disease; Glaucoma symptom scale
MeSH Terms: interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective laser trabeculoplasty (Experimental): Treating with the selective laser trabeculoplasty
  Interventions: Device: Selective laser trabeculoplasty
- Travoprost (Active Comparator): Using eye drop: travoprost
  Interventions: Drug: Travoprost

INTERVENTIONS:
Device: Selective laser trabeculoplasty — Selective laser trabeculoplasty platform The Lumenis Selecta® Duet™ (Lumenis Ltd., Yokneam, Israel)
  Other Names: The Lumenis Selecta® Duet™ (Lumenis Ltd., Yokneam, Israel)
  Arms: Selective laser trabeculoplasty
Drug: Travoprost — Travoprost benzalkonium-free ophthalmic solution (40 microgram/ml) (Alcon Laboratories, Inc., Fort Worth, TX, USA)
  Other Names: Travatan benzalkonium-free
  Arms: Travoprost

SUMMARY:
The investigators conduct this study to access the effect of selective laser trabeculoplasty on 24-hour circadian tension curves of patients with open-angle glaucoma, normal tension glaucoma and ocular hypertension. This treatment effect is compared with that of the prostaglandin analogue, travoprost.

DETAILED DESCRIPTION:
Selective laser trabeculoplasty is an effective treatment for lowering intraocular pressure in patients with open-angle glaucoma. Clinical evaluations of its effectiveness in individual patients usually are derived from baseline and post-laser measurements of intraocular pressure during office hours in the sitting position. Only a few studies have examined the efficacy of laser trabeculoplasty beyond office hours. Although the 24-hour effect of laser trabeculoplasty has been studied ,the study was conducted before the use of these new and more potent intraocular pressure lowering drugs. So it doesn't have any study to determine the effect of selective laser trabeculoplasty and travoprost to reduce the diurnal and nocturnal variation of Iintraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year-old
* Patients who were diagnosed as primary open-angle glaucoma, normal tension glaucoma, and ocular hypertension either newly diagnosed or currently on medical therapy.
* Agree to participate in the study, accept to be randomized to receive treatment, and willing to sign an informed consent

Exclusion Criteria:

Related to the severity of disease and visual acuity status

* Advance glaucoma in the study eye
* Have a very high intraocular pressure that need immediate treatment to prevent retinal vein occlusion (intraocular pressure >30 mmHg)
* Currently on maximal tolerated medical treatment and unable to control intraocular pressure
* Currently on oral carbonic anhydrase inhibitor for intraocular pressure control
* Single eye, the other eye blind from any cause

Related to surgical procedures

* Prior laser trabeculoplasty
* Prior glaucoma surgery
* Prior retinal surgery
* Underwent less than 3-month cataract extraction
* Potential need for other ocular surgery within the 2-3-month follow-up period since enrollment Related to underlying and ocular history
* History of diabetic retinopathy staged as severe non-proliferative or worse
* Narrow iridocorneal angle
* Ocular condition precluding visualization of trabecular meshwork
* Recently have ocular inflammation of any cause
* Previous history of ocular trauma
* Pregnant or breast-feeding women Related to the difficulty of having reliable measurements
* History of refractive surgery or any keratoplastic procedure
* Corneal opacities or diseases making no suitable tonometry
* Subjects with having poor or eccentric fixation or nystagmus
* Excessive eye squeezing
* Unable to lay down for measuring intraocular pressure in supine position during the night time
* Unable to have intraocular pressure checked every 2-hour such as have complicated underlying diseases or having sleep deprivation Related to allergy
* Known allergy to topical anesthesia
* Known allergy to fluorescein solution
* Known allergy to travoprost Related to compliance
* Impairment preventing adequate understanding to sign an informed consent
* Subject has demonstrated potential for non-compliance with the study protocol
* Unwilling to be randomized to receive treatment
* Unwilling to be washed out from currently treated drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of circadian intraocular pressure | Six weeks after recieving treatment
  intraocular pressure values measured during daytime and nighttime, compare between selective laser trabeculoplasty and travoprost (include pre- and post-treatment intraocular pressure values)

SECONDARY OUTCOMES:
Position related intraocular pressure | Six weeks after the treatments
  Intraocular pressure different when measuring in the sitting and supine position (include pre- and post-treatment intraocular pressure values
Ocular surface disease | Six weeks after the treatments
  Using the glaucoma symptom scale-10 (GSS-10) and ocular surface disease questionnaire for evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No